CLINICAL TRIAL: NCT03440112
Title: Modulation of GABA-A Receptors and Axial Motor Impairments in Parkinson
Brief Title: Modulation of GABA-A Receptors in Parkinson Disease-Transdermal Flumazenil Arm
Acronym: GABA-A
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nicolaas Bohnen, MD, PhD (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Nicolaas Bohnen, MD, PhD, Professor of Radiology and Neurology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HUM00360361-A; R01NS099535 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-20 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
Keywords: Gait; Balance; GABA; Transdermal flumazenil (previously Clarithromycin changed 4/2020); PET Imaging; MRI; Mobility
MeSH Terms: conditions — Parkinson Disease | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Clarithromycin (Not used anymore as of 4/2020; study aborted) (Active Comparator): Clarithromycin 250mg (1 capsule) will be taken orally twice a day for 3 days and if tolerated will be increased to 500mg (2 capsules) orally twice a day for 4-6 days.
  Interventions: Drug: Clarithromycin (Not used as of 4/2020)
- Placebo (Not used anymore as of 4/2020; study aborted) (Placebo Comparator): Placebo will be taken exactly as the clarithromycin arm: 1 capsule orally twice a day for 3 days and if tolerated will be increased to 2 capsules orally twice a day for 4-6 days.
  Interventions: Drug: Placebo (Not used as of 4/2020)
- Transdermal flumazenil (added 4/2020 as safer alternative for clarithromycin) (Active Comparator): Added in April 2020. Subjects will take 18mg transdermal application every 3-4 hrs dispensed as 3 dispenser bottle clicks of 0.25 ml each, while awake for 3 days then if no side-effects subjects will increase to 36mg transdermal application every 3-4 hrs dispensed as 6 dispenser bottle clicks of 0.25 ml each, while awake.
  Interventions: Drug: Transdermal flumazenil (Added 4/2020)
- Placebo cream (added 4/2020) (Placebo Comparator): Added in April 2020. Placebo will be taken exactly as the transdermal flumazenil arm: Subjects will take 18mg transdermal application every 3-4 hrs dispensed as 3 dispenser bottle clicks of 0.25 ml each, while awake for 3 days then if no side-effects subjects will increase to 36mg transdermal application every 3-4 hrs dispensed as 6 dispenser bottle clicks of 0.25 ml each, while awake.
  Interventions: Drug: Placebo (Added 4/2020)

INTERVENTIONS:
Drug: Clarithromycin (Not used as of 4/2020) — Clarithromycin (generic) capsule 250mg each
  Other Names: Biaxin
  Arms: Clarithromycin (Not used anymore as of 4/2020; study aborted)
Drug: Placebo (Not used as of 4/2020) — Lactose in a gel capsule
  Arms: Placebo (Not used anymore as of 4/2020; study aborted)
Drug: Transdermal flumazenil (Added 4/2020) — Transdermal flumazenil 24mg/mL
  Arms: Transdermal flumazenil (added 4/2020 as safer alternative for clarithromycin)
Drug: Placebo (Added 4/2020) — Transdermal placebo
  Other Names: Placebo cream
  Arms: Placebo cream (added 4/2020)

SUMMARY:
The arm of this study evaluates possible GABA-A receptor target engagement effects of the FDA-approved medication, transdermal flumazenil (added 4/2020, replaced clarithromycin), in the setting of Parkinson's disease. Half of the subjects will receive transdermal flumazenil for 7-10 days, and half will receive a placebo. [11C]Flumazenil GABA-A receptor PET imaging will be used to assess target engagement effects. Note [11C]Flumazenil GABA-A receptor PET was not performed as part of the transdermal flumazenil study because of a Covid pandemic research amendment.

DETAILED DESCRIPTION:
This study focuses on neurochemical changes in the brain that occur in Parkinson's disease. In particular we will be looking a neurotransmitter called GABA. In some Parkinson's disease patients we see too much GABA activity in the brain. This target engagement study examines the target engagement effect of GABA-A receptor modulation by transdermal flumazenil (previously clarithromycin). [11C]-flumazenil Positron Emission Tomography (PET) imaging results will be used to assess for possible GABA-A receptor target engagement effects of transdermal flumazenil (previously clarithromycin). Note [11C]Flumazenil GABA-A receptor PET was not performed as part of the transdermal flumazenil study because of a Covid pandemic research amendment.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease (PD): PD diagnosis will follow the UK Parkinson's Disease Society Brain Bank Research Center (UKPDSBRC) clinical diagnostic criteria for PD.
2. Hoehn and Yahr stages 2-4
3. Absence of dementia confirmed by cognitive testing.
4. Abnormal 11C-Dihydrotetrabenazine ([11c]-DTBZ) PET study to demonstrate nigrostriatal dopaminergic denervation

Exclusion Criteria:

1. PD with Dementia (PDD) or dementia with Lewy bodies (DLB).
2. Other disorders which may resemble PD, such as vascu¬lar dementia, normal pressure hydrocephalus, multiple system atrophy, corticobasal ganglionic dege¬neration, or toxic causes of parkinsonism. Prototypical cases have distincti¬ve clinical profiles, like early and severe dysautonomia or appendicular apraxia, which may differentiate them from idiopathic PD. The use of the UKPDSBRC clinical diagnostic criteria for PD will mitigate the inclusion of subjects with atypical parkinsonism.
3. Subjects currently on benzodiazepine, GABAB-ergic medications (baclofen, tizanidine), modafinil, neuroleptic, anticholinergic (trihexyphenidyl, benztropine), or cholinesterase inhibitor drugs.
4. Evidence of a mass lesion on structural brain imaging (MRI).
5. Participants in whom MRI is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, chest, or cochlear implant.
6. Severe claustrophobia precluding MR or PET imaging.
7. Subjects limited by participation in research procedures involving ionizing radiation.
8. Pregnancy (urine or serum pregnancy test within 48 hours of each PET session) or breastfeeding.
9. History of seizures
10. Significant anxiety or history of panic disorder.
11. History of recent suicide attempt or overdose of tricyclic antidepressants or other medications.
12. History of transient ischemic attack (TIA) or stroke within the last year.
13. History of systemic lupus erythematosis.
14. Abnormal liver enzymes (AST or ALT) > 3 times upper limit of normal.
15. History of atrial fibrillation.
16. History of retinal branch artery occlusion.
17. Active dermatitis inner forearms.
18. Any other medical history determined by investigators to preclude safe participation.

Additional Exclusion Criteria for Flumazenil sub-studies:

1. Allergy to flumazenil
2. Significant liver disease
3. History of alcohol or other substance abuse within past two years.
4. Subjects currently taking benzodiazepines

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas I Bohnen, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System Functional Neuroimaging, Cognitive and Mobility Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants withdrew prior to assignment. 7 participants were recruited for clarithromycin sub-study, which was subsequently dropped in 04/2020 due to concerns related to increased risk of death among the elderly who were taking this antibiotic even for a short time. Only 3 of those participants were randomized and went through study procedures, but the randomization key was not broken so we have no way of knowing what group they were assigned to.
Groups:
- Transdermal Flumazenil (Active): Subjects will take 18mg transdermal application every 3-4 hrs dispensed as 3 dispenser bottle clicks of 0.25 ml each, while awake for 3 days then if no side-effects subjects will increase to 36mg transdermal application every 3-4 hrs dispensed as 6 dispenser bottle clicks of 0.25 ml each, while awake.
- Placebo Cream: Placebo will be taken exactly as the transdermal flumazenil arm: Subjects will take 18mg transdermal application every 3-4 hrs dispensed as 3 dispenser bottle clicks of 0.25 ml each, while awake for 3 days then if no side-effects subjects will increase to 36mg transdermal application every 3-4 hrs dispensed as 6 dispenser bottle clicks of 0.25 ml each, while awake.
- Oral Clarithromycin (Dropped in 04/2020): Subjects will take 250 mg twice daily by mouth for 3 days and then - if no side-effects - the dose will increased to 500 mg twice daily by mouth.
Period: Overall Study
Arm/Group | Transdermal Flumazenil (Active) | Placebo Cream | Oral Clarithromycin (Dropped in 04/2020)
Started | 11 | 11 | 3
Completed | 11 | 11 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Parkinson's disease patients age 50 years or older. Some, but not all, participants in the Clarithromycin arm were randomized, and only few completed study procedures because of premature termination of the trial due to an FDA safety risk warning of Clarithromycin, precluding any meaningful analysis. Consequently, this study arm was replaced by the transdermal Flumazenil arm.
Groups:
- Transdermal Flumazenil (Active): Added in April 2020. Subjects will take 18mg transdermal application every 3-4 hrs dispensed as 3 dispenser bottle clicks of 0.25 ml each, while awake for 3 days then if no side-effects subjects will increase to 36mg transdermal application every 3-4 hrs dispensed as 6 dispenser bottle clicks of 0.25 ml each, while awake.
- Placebo Cream: Added in April 2020. Placebo will be taken exactly as the transdermal flumazenil arm: Subjects will take 18mg transdermal application every 3-4 hrs dispensed as 3 dispenser bottle clicks of 0.25 ml each, while awake for 3 days then if no side-effects subjects will increase to 36mg transdermal application every 3-4 hrs dispensed as 6 dispenser bottle clicks of 0.25 ml each, while awake.
- Oral Clarithromycin (Active or Placebo): Discontinued April 2020, study aborted. Subjects will take 250 mg twice daily by mouth for 3 days and then - if no side-effects - the dose will increased to 500 mg twice daily by mouth.
- Total: Total of all reporting groups
Arm/Group | Transdermal Flumazenil (Active) | Placebo Cream | Oral Clarithromycin (Active or Placebo) | Total
Number analyzed (Participants) | 11 | 11 | 3 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.09 (4.41) | 70.27 (3.80) | 66.33 (5.13) | 70.6 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 8 | 10 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 3 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 11 | 3 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 3 | 25
MiniBEST Sensory Subscore [Mean (Standard Deviation); unit: units on a scale] — MiniBEST sensory subscore measures an individual's ability to maintain balance under conditions of sensory constrain and unstable/inclined standing surface. It is is computed as a sum of MiniBEST items 7, 8, and 9.The score ranges from 0 to 6, with 0 indicating inability to balance under all of the condition, and 6 indicating no difficulty in maintaining balance under any of the conditions (lower score indicates worse balance). Baseline measure was collected during pre-clinical screening visit in dopaminergic medication OFF state.
  units on a scale | 5.27 (1.1) | 5.81 (0.40) | 6 (0) | 5.6 (0.82)
Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III [Median (Inter-Quartile Range); unit: units on a scale] — We will use the total Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III - motor scale to assess motor function. Scale from 0-132, higher scores indicate worse motor outcomes. Baseline measure was collected during pre-clinical screening visit in dopaminergic medication OFF state.
  units on a scale | 45 [38.5 to 57] | 41.5 [37 to 49.25] | 40.50 [33.00 to 45.25] | 43.5 [36.00 to 51.50]

OUTCOME MEASURES:

1. Primary Outcome: Change in Quantitative Biomechanics 1 (Clinical Motor Ratings MDS-UPDRS)
Description: We will use the total Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III - motor scale rating scores to assess motor function. Scale from 0-132, higher scores indicate worse motor outcomes. Outcome measure was collected during dopaminergic medication ON state.
Time Frame: Day 1 (before treatment administration), day 7 (after 7 days of treatment), and day 14 (7 days of treatment discontinuation).
Population: Parkinson's disease participants older than 50. Some, but not all, participants in the Clarithromycin arm were randomized, and only few completed study procedures because of premature termination of the trial due to an FDA safety risk warning of Clarithromycin, precluding any meaningful analysis. Consequently, this study arm was replaced by the transdermal Flumazenil arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Clarithromycin (Active or Placebo): Discontinued April 2020. Subjects will take 250 mg twice daily by mouth for 3 days and then - if no side-effects - the dose will increased to 500 mg twice daily by mouth.
Arm/Group | Transdermal Flumazenil (Active) | Placebo Cream | Clarithromycin (Active or Placebo)
Number analyzed (Participants) | 11 | 11 | 3
units on a scale
  Day 1 | 38 [27.5 to 44.5] | 34 [30 to 47] | 28 [25.50 to 33.00]
  Day 7 | 36.75 [29.75 to 52] | 31.50 [25.375 to 43.375] | 23.50 [21.25 to 26.75]
  Day 14 | 32.75 [26.375 to 47.375] | 34 [29.5 to 40] | 22 [19.5 to 23.0]
Statistical Analysis 1: Comparison: Transdermal Flumazenil (Active) vs Placebo Cream; A pair of random-intercept mixed linear models was fitted, a visit model and an interaction model. Visit model included fixed effect of visit and a random intercept by participant. Interaction model adds an interaction by treatment term on top of the visit model. Null hypothesis is that visit by treatment interaction does not explain significant additional variance in clinical outcome scores. Likelihood ratio test comparing the interaction model to the visit model was used to derive a p-value; Test type: Superiority; p = 0.391, Mixed Models Analysis; Chi-Squared = 3.0039

2. Secondary Outcome: Change in Quantitative Biomechanics 2 (MiniBESTest Dynamic Balance Scale Sensory Subscore)
Description: MiniBEST sensory subscore measures an individual's ability to maintain balance under conditions of sensory constrain and unstable/inclined standing surface. It is is computed as a sum of MiniBEST items 7, 8, and 9.The score ranges from 0 to 6, with 0 indicating inability to balance under all of the condition, and 6 indicating no difficulty in maintaining balance under any of the conditions (lower score indicates worse balance). Outcome measure was collected during dopaminergic medication ON state.
Time Frame: as for outcome 1
Population: Parkinson's disease participants older than 50. Some, but not all, participants in the Clarithromycin arm were randomized, and only few completed study procedures (baseline visit only) because of premature termination of the trial due to an FDA safety risk warning of Clarithromycin, precluding any meaningful analysis. Consequently, this study arm was replaced by the transdermal Flumazenil arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Clarithromycin (Active or Placebo): Discontinued April 2020. Subjects will take 250 mg twice daily by mouth for 3 days and then - if no side-effects - the dose will increase to 500 mg twice daily by mouth.
Arm/Group | Transdermal Flumazenil (Active) | Placebo Cream | Clarithromycin (Active or Placebo)
Number analyzed (Participants) | 11 | 11 | 3
units on a scale
  Day 1 | 5.54 (0.69) | 6 (0) | 6 (0)
  Day 7 | 5.82 (0.40) | 6 (0) | 5.67 (0.58)
  Day 14 | 6 (0) | 5.82 (0.60) | 6 (0)
Statistical Analysis 1: Comparison: Transdermal Flumazenil (Active) vs Placebo Cream; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.02351, Mixed Models Analysis; Chi-Squared = 9.4836

ADVERSE EVENTS:
Time Frame: Up to 14 days.
Arm/Group | Transdermal Flumazenil (Active) | Placebo Cream | Oral Clarithromycin (Dropped in 04/2020)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/3

LIMITATIONS AND CAVEATS:
Our participants were predominantly male, which is often the case with Parkinson's disease (PD) patient population since PD is known to affect males at a greater rate. This means that our findings may not generalize as well to population of female PD patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT03440112/Prot_003.pdf
  • Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03440112/SAP_004.pdf